CLINICAL TRIAL: NCT00070746
Title: Perinatal Infections and Pregnancy Outcomes in Pakistan: A Collaborative Research Project in Partnership With the University of Alabama, USA
Brief Title: Perinatal Infections in Pakistan
Status: Completed | Type: Observational
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); University of Alabama at Birmingham (Other); Aga Khan University (Other)
Responsible Party: Sponsor
Other Study IDs: GN 09; U01HD040607 (NIH)
Record Dates: First submitted 2003-10-07; First posted 2003-10-10 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Bacterial Vaginosis; Fetal Membranes, Premature Rupture; Chorioamnionitis; Pregnancy
Keywords: Perinatal mortality [PNM]; Neonatal mortality; Low birth weight [LBW]; Spontaneous preterm delivery [SPTD]; Premature rupture of membranes [PROM]; Histological chorioamnionitis; Global Network; Pakistan; Maternal and child health; International; Women's health
MeSH Terms: conditions — Vaginosis, Bacterial; Fetal Membranes, Premature Rupture; Chorioamnionitis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There are large differences in health outcomes related to pregnancy and birth between developed and developing countries. This study will investigate how infections, medical history, health care behavior and psychosocial issues are associated with pregnancy outcomes in Pakistan.

DETAILED DESCRIPTION:
Pakistan, the world's seventh most populous country of about 138 million people, is beset with severe problems in its maternal and child health sector. The official maternal mortality ratio for Pakistan is reported as 340 per 100,000 live births.

The overall goal to conduct a prospective observational study to identify the risk factors for adverse pregnancy outcomes including reproductive tract infections such as BV, and other physical, dental, nutritional, psychosocial, and behavioral characteristics. The primary objective is to examine the association between BV in pregnant women at 20-26 weeks gestation and various other biochemical infection markers with adverse pregnancy outcomes (i.e., perinatal mortality [PNM], neonatal mortality, low birth weight [LBW], spontaneous preterm delivery [SPTD], premature rupture of membranes [PROM], histological chorioamnionitis).

Additionally, this study will explore the relationship of various health behaviors and health status to the presence of perinatal infections. A total of 1,500 pregnant women will be enrolled in the study. A matched case-control study will be conducted at the end of the data collection period to evaluate the use of markers for the prediction of infection related perinatal mortality and infection related SPTD. All investigators and laboratory personnel will remain blinded to the identity of specimens through the use of unique study identifier numbers. Collected data will then be unblinded, analysed, and correlated with the previously collected demographic, obstetrics, and neonatal outcome, microbiology and histopathological data.

Based on the findings of this study, appropriate interventions to address reproductive tract infection (RTI) could be developed and field-tested in Pakistan. We expect that these interventions, once successfully field-tested, could be widely used to improve maternal and child survival in Pakistan and other developing countries. Given the critical state of maternal and child health in Pakistan, and considering the emerging evidence that infections could lead to poor pregnancy outcomes, this study is extremely relevant and timely, and it has the potential to contribute significantly toward the improvement of reproductive health in Pakistan. Primary outcome is perinatal mortality. Secondary outcomes include birth weight; spontaneous delivery occurring before 37 weeks gestation; rupture of fetal membranes before 37 weeks of gestation; and maternal death. The sample size was based on 25% prevalence of BV in the control group; 10 percent dropout rate; 80 percent power; and a two-tailed type I error of 0.05.

ELIGIBILITY:
Inclusion Criteria:

Participants must

* be in their 20th to 26th week of pregnancy (to be confirmed by an ultrasound)
* be permanent residents (resident for the past months or intending to stay for next the 6 months) of the study site in Hyderabad, Pakistan; and,
* give informed (written or verbal) consent.

Exclusion criteria:

* have clinical diagnoses of life-threatening conditions (requiring immediate treatment or hospitalization, as diagnosed by the attending physician).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 2003-06; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Robert Goldenberg, MD, Principal Investigator — Drexel University
Locations (1):
- Health clinic, Hyderābād, Pakistan

REFERENCES:
- See also: Website for the Global Network for Women's and Children's Health Research. — http://gn.rti.org
- See also: Research Triangle Institute International — http://www.rti.org
- See also: Aga Khan University, Pakistan — http://www.aku.edu/